CLINICAL TRIAL: NCT06788041
Title: ANALYSIS OF THE EFFECT OF HAMMAM EXPERIENCE ON GENERAL HEALTH AND PERCEIVED WELL-BEING COMPARED TO MASSAGE AND PLACEBO : A RANDOMIZED CROSS-SECTIONAL STUDY.
Brief Title: EFFECT OF HAMMAM EXPERIENCE ON GENERAL HEALTH AND PERCEIVED WELL-BEING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: AL ÁNDALUS BAÑOS ÁRABES (Hammam Granada) (Unknown)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, Professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: HAM24
Record Dates: First submitted 2024-12-07; First posted 2025-01-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Stress; Wellness; General Health
Keywords: hamman; balneotherapy; massage; chronic stress; general health; wellness
MeSH Terms: interventions — Balneology; Massage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 (ABC) (Experimental): Participants in this arm will rotate through three treatments (Treatment A Hamman experience and massage, Treatment B massage only, and Treatment C placebo) in a randomized sequence. Each treatment will be separated by a washout period to minimize carryover effects. All participants will experience each treatment at different periods, serving as their own control.
  Interventions: Other: Hamman experience; Other: Massage; Other: Placebo Comparator
- Arm 2 (ACB) (Experimental)
  Interventions: Other: Hamman experience; Other: Massage; Other: Placebo Comparator
- ARM 3 (BAC) (Experimental)
  Interventions: Other: Hamman experience; Other: Massage; Other: Placebo Comparator
- Arm 4 (BCA) (Experimental)
  Interventions: Other: Hamman experience; Other: Massage; Other: Placebo Comparator
- Arm 5 (CAB) (Experimental)
  Interventions: Other: Hamman experience; Other: Massage; Other: Placebo Comparator
- Arm 6 (CBA) (Experimental)
  Interventions: Other: Hamman experience; Other: Massage; Other: Placebo Comparator

INTERVENTIONS:
Other: Hamman experience — There will be a circuit in the Hammam Al Andalus baths with baths in all pools (warm, hot or cold water) and sauna for 30 minutes. The time in each pool will be determined by the sensation and tolerance of each participant. In addition, participants will receive foam with aromatic oils on the participant's body (arms, trunk and legs). This foam will be left for about 10 minutes on the participant's body, while a manual body therapy is performed. The force to be applied will be very weak, a superficial rubbing will be performed to prepare the tissue, followed by a maintained pressure and then sliding pressures are performed. The application time should not exceed 15 minutes.
  Other Names: Balneotherapy and massage
Other: Massage — Duration of 45 minutes. A complete dorsal and ventral body massage will be performed, with superficial maneuvers at a slow pace of traditional massage.
Other: Placebo Comparator — The person will be instructed to stay for 45 minutes during which he/she will receive different electrotherapy techniques with the devices disconnected, a mobile device that simulates a beep will be placed so that the patient believes that the device is connected.

SUMMARY:
The main objective of this study is to analyze the effect of a Hammam experience, a massage experience and a placebo in a healthy general population on their general health and perception of well-being, assessed with biophysiological, physical and psychoemotional markers, and its impact on chronic stress. Our hypothesis is that the Hammam experience will produce a more favorable acute (just after the experience) and subacute (24 hours after the experience) response on the study variables than the other interventions with at least a moderate effect size.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (50%) 25-65 years old
* No metabolic risk.
* Resident in the province of Granada.
* Socio-economic level: medium-high
* Experience in self-care
* Spanish level C2

Exclusion Criteria:

* Pregnancy
* Participation in treatments and relaxation techniques or taking medication (anxiolytics) frequently (≥ 1 per week) in the last 12 months
* Medical situations limiting participation in the study: acute musculoskeletal pathologies (fractures, wounds, etc.) or local inflammatory processes, diagnosed psychiatric disease, vascular diseases (thrombosis), contagious diseases, fever, thermoregulation problems, incontinence, craniocerebral trauma or infarction (< 6 months), thermal allergies, hypertension, or any uncontrolled systemic disease).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Balance of the autonomic nervous system upon waking | Measurement 1: Upon waking on the session day (6:00-7:00 a.m.); Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 4: Upon waking the day after session (6:00-7:00 a.m.); Measurement 5: 2
  Evaluated through heart rate variability upon waking up. It will always be performed under the same conditions in an unlit, quiet environment without noise/distractions, with the person in supine position and after emptying the bladder. A total time of 5 min will be recorded through H-10 polar band.

SECONDARY OUTCOMES:
Sleep satisfaction | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Assessed through a Likert scale in which 0 corresponds to the option "Not all all satisfactory" and 10 with "Very satisfactory"
Hours of sleep | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Assessed through an open question in which participants are asked "What time did you go to bed to sleep?", "What time did you wake up in the morning?" and "How many hours and minutes do you think you slept in total at night?"
Perception of well-being | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Assessed with the EBS-8 subjective well-being scale, which assesses the two components of well-being: life satisfaction and positive affect and with a visual analog scale 0-10.
Mood | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  The Mood Rating Scale (EVEA) will be used, which evaluates mood states with a range from 0 to 10 and as a time reference "right now". It consists of 4 subscales: sadness-depression, anxiety, anger-hostility and joy.
Mental agility | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Assessed by the "Trail Marking Test", which assesses t used to evaluate attention, flexibility of thought and visuospatial ability. It consists of two parts. In both cases, the subject will need a pencil and the evaluator a stopwatch, counting the execution time for each of the parts as soon as the pertinent indications have been given. In part A, the participant will join in ascending order all the numbers from 1 to 25 arranged on a sheet of paper. In exercise B, the process will be repeated, but alternating letters and numbers in alphanumeric order. In both cases, the time spent will be quantified.
Distress | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Assessed through a distress thermometer, a likert scale in which 0 corresponds to the option "No distress" and 10 with "Extreme distress"
Flexibility | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  The "sit and reach" test will be performed, for the evaluation of flexibility in which the subject, who is seated on the edge of a chair (placed against a wall for safety reasons), and one foot resting on the sleep, will extend the other leg forward with the knee straight, the heel resting on the sleep and the ankle at 90º, placing one hand on top of the other with the tips of the central fingers equal. The participant will be instructed to inhale and, on exhalation, extend the hand forward toward the toes by bending at the hip. The distance will be measured between the fingertips and toes so that, if the fingertips touch the toes, the score is 0, if they do not touch, the resulting distance in cm will be negative and, if they overlap, we are talking about a distance in cm positive.
Functional capacity | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  With the sit-to-stand test 30 seconds, which measures how many times a person can transition from sitting in a chair to standing and back to sitting within 30 seconds.
Fatigue | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  After completing the 30-second sit-to-stand test, participants rate their perceived level of fatigue using the Borg CR10 scale. This scale ranges from 0 (no fatigue at all) to 10 (extreme fatigue) and provides a subjective measure of exertion following the activity.
Overall stress regulation | Measurement 1: Upon waking on the session day (6:00-7:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 4: Upon waking the day after session (6:00-7:00 a.m.).
  Salivary samples will be collected first thing in the morning, using a timer and ensuring the entire sample is collected within three minutes. Without ingestion of caffeine and/or stimulant substances 12 hours before, as well as with complete oral hygiene (dental brushing and use of mouthwash, preferably) the night before.
  Salivary samples (400µL) will be collected in specific collection kits for 2ml salivary sample and cryovials (Salimetrics, LLC, Carlsbad, United States), to proceed to their subsequent immediate freezing at -80ºC until the pertinent analysis of cortisol through ELISA is performed.
Systolic blood pressure | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Measured with the patient seated after at least 10 minutes of rest using a sphygmomanometer.
Diastolic blood pressure | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Measured with the patient seated after at least 10 minutes of rest using a sphygmomanometer.
Heart rate | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Measured with the patient seated after at least 10 minutes of rest using a sphygmomanometer
Blood oxygen saturation | Measurement 2: 30 minutes before session (8:00 a.m.); Measurement 3: 5 minutes after session (10:00 a.m.); Measurement 5: 24 hours post-session (8:00 a.m.).
  Measured using a pulse oximeter placed on the fingertip, ensuring the patient is seated and at rest for at least 10 minutes prior to measurement.

OTHER OUTCOMES:
Attitude and beliefs towards holistic treatment | Measurement 0: At enrollment
  Through the Complementary and Alternative Medicine Health Belief Questionnaire (CHBQ), validated to Spanish.It has 10 items and addresses perception of the effectiveness of alternative therapies; willingness to use holistic treatments; and trust in complementary medicine practitioners.
Previous experience participating in holistic therapeutic modalities. | Measurement 0: At enrollment
  Assessed through a yes/no questionnaire to determine prior experiences, followed by an open-ended question to record the type of modality if applicable
Level of perceived stress | Measurement 0: At enrollment
  The Perceived Stress Scale (PSS-10) is a self-assessment tool used to measure the level of perceived stress in individuals in his or her life during the past month. The scale consists of 10 questions that explore different aspects of perceived stress, such as how often individuals feel that their life is out of control, feel nervousness, or are unable to cope with their responsibilities. The total score is obtained by summing the item responses. Some questions are positively worded and are reverse scored.
Resilience | Measurement 0: At enrollment
  The Connor-Davidson Resilience Scale (CD-RISC) is a self-assessment tool that measures a person's ability to overcome adversity. It is composed of 25 items that are answered on a 5-point Likert scale, ranging from 0 (never) to 4 (almost always). Total scores can range from 0 to 100, with higher scores indicating greater resilience.
Age | Measurement 0: At enrollment
  Will be collected using an open-ended questionnaire where participants will provide their exact age
Place of Residence | Measurement 0: At enrollment
  Will be collected using an open-ended questionnaire where participants will provide their Place of Residence
Employment status | Measurement 0: At enrollment
  Will be assessed through a multiple-choice questionnaire, allowing participants to select the most appropriate response for their situation.
Marital Status | Measurement 0: At enrollment
  Will be assessed through a multiple-choice questionnaire, allowing participants to select the most appropriate response for their situation.
Level of Education | Measurement 0: At enrollment
  Will be assessed through a multiple-choice questionnaire, allowing participants to select the most appropriate response for their situation.
Family Income | Measurement 0: At enrollment
  Will be collected using a range-based question, where participants will indicate the income bracket that best reflects their household's monthly or annual income
Height | Measurement 0: At enrollment
  Measured using a calibrated stadiometer with participants standing upright and barefoot
Weight | Measurement 0: At enrollment
  Measured using digital scale, with participants standing barefoot, and in light clothing.
Waist Circumference | Measurement 0: At enrollment
  Measured using a non-stretchable tape, ensuring standard anatomical landmarks are used: between last ribs and iliac creast, at the narrowest point
Hip Circumference | Measurement 0: At enrollment
  Measured using a non-stretchable tape, ensuring standard anatomical landmarks are used: above the greater trochanter
Waist-Hip Ratio | Measurement 0: At enrollment
  Calculated by dividing waist circumference by hip circumference
Drug consumption | Measurement 0: At enrollment
  These behaviors will be assessed through a structured questionnaire, including frequency and quantity of use over the past months.
Sedentary Behavior | Measurement 0: At enrollment
  Measured using questions about time spent sitting or reclining during typical weekdays and weekends, excluding sleep hours
Physical Activity Levels | Measurement 0: At enrollment
  Physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ), which captures the type, frequency, and duration of physical activities performed weekly, categorized into light, moderate, and vigorous intensity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided